CLINICAL TRIAL: NCT06231472
Title: Preemptive Weight-Based Fluid Therapy Reduces Post-Induction Hypotension in Gynecological Pelvic Surgery: A Randomized Controlled Trial Using IVC Ultrasonography
Brief Title: Effect of Preoperative Fluid Therapy on Post-induction Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Burgac (Other)
Responsible Party: Sponsor-Investigator, Mustafa Burgac, chief researcher, Assistant doctor, Istanbul Medeniyet University
Organization: Istanbul Medeniyet University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022/0263
Record Dates: First submitted 2023-12-22; First posted 2024-01-30 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hypovolemia
Keywords: Post-induction hypotension, Preemptive fluid therapy
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Intervention Model Description: In the preoperative period, two groups were created: patients who received weight-based fluid therapy and patients who did not receive weight-based fluid therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A with preoperative weight-based fluid therapy (Other): Group A patients received fluid infusion calculated according to hourly weight before surgery.
  Interventions: Other: weight-based fluid therapy
- Group B without preoperative weight-based fluid therapy (No Intervention): No intervention was made to patients in group B.

INTERVENTIONS:
Other: weight-based fluid therapy — Group A received weight-based fluid therapy throughout the preoperative fasting period, whereas Group B did not receive any preoperative treatment.
  Arms: Group A with preoperative weight-based fluid therapy

SUMMARY:
Although preoperative dehydration is a known risk factor for post-induction hypotension, evidence regarding preemptive weight-based fluid therapy remains limited. This study aimed to assess whether preemptive weight-based fluid therapy during fasting reduces the risk of post-induction hypotension.

This trial randomized 122 patients. After excluding 12 patients (10 for non-visualized IVC, 2 for vasoactive agents), 110 patients (55 per group) were analyzed. Group A received preemptive fluid therapy versus Group B's standard fasting. The primary objective of the study was to evaluate the efficacy of preemptive weight-based fluid therapy on the prevention of post-induction hypotension following general anesthesia (Mean blood pressure/MBP < 60 mmHg or ≥ 30% decrease from baseline). Secondary outcomes included ultrasonographic parameters (Inferior vena cava diameter/dIVC, collapsibility index/CI%) and hemodynamic indices (Perfusion index/PI, pleth variability index/PVI, pulse pressure variation/PPV). Statistical analyses included receiver operating characteristic (ROC) curves and logistic regression.

DETAILED DESCRIPTION:
This prospective, randomized, controlled study was approved by the Ministry of Health, Istanbul Medeniyet University, Göztepe Training and Research Hospital Clinical Research Ethics Committee (approval number 2022/0263, dated 27 April 2022) and was registered in ClinicalTrials.gov (NCT 06231472). The study was conducted by the principles outlined in the Declaration of Helsinki. Written and verbal informed consent was obtained from all participants.

This study was conducted between May 2022 and November 2023. A total of 122 female patients aged 18 years and older, scheduled for gynaecological pelvic surgery with an American Society of Anaesthesiologists (ASA) physical status score of I-III, were included in this study. Exclusion criteria included unstable haemodynamics (persistent hypotension preventing extubation, arrhythmia, ejection fraction/EF < 40%), valvular heart disease, cardiac pacing, obesity (Body mass index/BMI >35), chronic obstructive pulmonary disease (COPD), increased intra-abdominal pressure, open wounds at the ultrasound site, preoperative severe hypertension (systolic blood pressure/SBP > 180 mmHg, diastolic blood pressure/DBP > 110 mmHg), use of angiotensin II receptor blockers (ARB), angiotensin-converting enzyme inhibitors (ACE-I), and refusal to participate in the study.

Randomization was performed using the sealed envelope method. Envelopes were randomly numbered, and each patient selected an envelope to determine her group. Patients who selected an envelope with an even number were assigned to Group A (n = 55), while those who selected an envelope with an odd number were assigned to Group B (n = 55).

All patients underwent preoperative evaluation and medical optimization in the preoperative assessment clinic. A detailed explanation of the weight-based fluid therapy protocol was provided to the patients on the evening before surgery, and informed consent was obtained. Bowel preparation was performed by the gynecological surgery team, and oral intake was discontinued at midnight in accordance with standard institutional protocols.

Patients in Group A were managed according to a weight-based intravenous fluid protocol. The fluid was administered during the preoperative fasting period using a standardized formula: 4 mL/kg for the first 10 kg of body weight, 2 mL/kg for the next 10 kg, and 1 mL/kg for each remaining kilogram. Patients in Group B, who served as the control group, did not receive any preoperative fluid therapy. The total volume of fluid administered to Group A was calculated and documented upon the patient's arrival in the operating room.

Once in the operating theatre, standard monitoring was initiated, including 5-lead electrocardiography (ECG), pulse oximetry, and non-invasive blood pressure monitoring (Fabius GS Premium Drager Anesthesia monitor). A Masimo Rainbow (Adult/Neonatal Pulse CO-Oximeter Adhesive sensor) probe was placed on the left index finger for the measurement of PI and PVI.

Preoperative US assessment of the IVC was performed while the patient was spontaneously breathing in the supine position for at least 5 minutes before induction [14]. The IVC was visualized using a low-frequency convex probe (CA1-7AD Samsung probe) under a subcostal approach with the US (Samsung Medison H60 system). The maximum (IVC max) and minimum (IVC min) diameters of the IVC were measured during the respiratory cycle, and the CI (%) was calculated using the formula:

CI (%) = (dIVCexp-dIVCinsp) / dIVCexp ×100 Where dIVC_exp is the expiratory diameter, and dIVC_insp is the inspiratory diameter of the IVC.

For anesthesia induction, 1 mg/kg midazolam and 1 µg/kg fentanyl were administered intravenously for sedation. Induction agents included 2 mg/kg propofol and 0.6 mg/kg rocuronium bromide. Anesthesia maintenance was achieved using a sevoflurane/oxygen/air mixture with a minimum alveolar concentration (MAC) of 0.8-1.0, and remifentanil was infused at 0.05-1 µg/kg/min as an analgesic. Ventilation settings included a tidal volume of 8 ml/kg, a frequency of 12-16 breaths/min, and positive end-expiratory pressure (PEEP) of 5 cm/H2O.

After induction, an intravenous cannula was inserted into the right radial artery under aseptic conditions for invasive blood pressure monitoring. PPV was recorded post-induction. Non-invasive measurements of heart rate (HR), SBP, MBP, PI, PVI, and PPV were recorded every 10 minutes during the intraoperative period.

Hypotension was defined as an MBP < 60 mmHg or a decrease of 30% or more from baseline. Patients who developed hypotension (Group H) were treated with a 3 ml/kg bolus of infused fluid, and IV 5 mg ephedrine was administered if haemodynamics did not improve. Fluid replacement was provided according to the surgical fluid losses and diuresis during the intraoperative period.

Anaesthesia was discontinued at the end of surgery. Neuromuscular blockade was reversed using IV sugammadex. Patients who met extubation criteria were transferred to the recovery room and later discharged to the ward after achieving a Modified Aldrete score of 12.

The primary outcome of this study was to compare the incidence of hypotension following anaesthesia induction between two groups of patients undergoing elective pelvic gynecological surgery with mechanical bowel preparation: patients receiving prophylactic weight-based fluid therapy (Group A) and those who did not (Group B). Secondary outcomes included the assessment of the predictive efficacy of dIVC, CI (%), PI, PVI, and PPV parameters for hypotension in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Gynaecological pelvic surgery planned for patients aged 18 years and over
* Patients with an American Society of Anaesthetists score of 1-2-3

Exclusion Criteria:

* Unstable haemodynamics (persistent hypotension preventing extubation at the end of surgery, arrhythmia, ejection fraction (EF) < 40%),
* Valvular heart disease,
* Cardiac pacing,
* Obesity (BMI >35),
* Chronic obstructive pulmonary disease (COPD),
* Increased intrabdominal pressure,
* Open wound at the US site,
* Preoperative severe hypertension (systolic blood pressure >180 mmHg, diastolic >110 mmHg),
* Use of angiotensin II receptor blockers (ARB), angiotensin coverting enzyme inhibitor (ACE-I)
* Refusal to participate in the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome was a comparison of the incidence of post-induction hypotension between the two groups. | perioperative/procedural
  All patients were thoroughly evaluated and medically optimised through the preoperative preparation outpatient clinic. The procedure for intra venous (IV) fluid infusion calculated according to preoperative weight was explained to the patient on the night of surgery and consent was obtained. Bowel cleansing procedure was performed by the gynaecological surgeon. Oral nutrition was discontinued at midnight, adhering to the routine practice of the gynaecology clinic. In Group A patients, maintenance fluid infusion calculated according to weight was started IV. The maintenance fluid calculated according to weight was infused hourly during the fasting period according to the method of 4 mL/st for the first 10 kg, 2 mL/st for the second 10 kg and 1 mL/st for each remaining kg.

SECONDARY OUTCOMES:
Secondary outcomes included the effect of PI, and PVI (%) in predicting hypotension. | perioperative/procedural
  Baseline measurements of PI and PVİ (%) were recorded before induction of general anaesthesia. PI, and PVI (%) measurements were recorded every 10 minute throughout the procedure. PVI (%) = [(PI max - PI min) / PI max] x 100 calculated with the formula. Measurements were recorded every 10 minutes throughout the procedure
Secondary outcomes included the effect of dIVC mm in predicting hypotension. | perioperative/procedural
  IVC ultrasonography was performed before induction. The IVC was visualised in M-mode using a subcostal approach from its junction with the right atrium on the paramedian long axis. Minimum and maximum inferior vena cava diameters (millimetres) due to respiratory cycle were measured in M-mode.
Secondary outcomes included the effect of PPV in predicting hypotension. | perioperative/procedural
  Baseline measurements of PPV were recorded after induction of general anaesthesia. PPV measurements were recorded every 10 minute throughout the procedure. PPV= (PPmaks-PPmin)/PPort. x 100 calculated with the formula. Measurements were recorded every 10 minutes throughout the procedure
Secondary outcomes included the effect of CI (%) in predicting hypotension. | perioperative/procedural
  Minimum and maximum inferior vena cava diameters (millimetres) due to respiratory cycle were measured in M-mode. The inferior vena cava collapsibility index (IVC-CI)= (dIVC expiration-dIVC inspiration) × 100/dIVCexpiration was calculated using the formula and recorded as a percentage. Measurements were recorded every 10 min throughout the procedure

CONTACTS AND LOCATIONS:
Overall Officials: hasan koçoğlu, Study Director — clinic chief
Locations (1):
- Istanbul Professor Doctor Süleyman Yalçın City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants' personal information will not be shared. Only the data and results used during the Study will be disclosed.